CLINICAL TRIAL: NCT05306145
Title: A Prospective, Single-center, Randomized Controlled Trial Comparing the Efficacy and Safety of High Freqnence Irreversible Electroporation and Trans Urethral Resection Prostate for Benign Prostatic Hyperplasia
Brief Title: Comparison of H-FIRE and TURP in Treating Benign Prostatic Hyperplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-FIREBPH-2021001
Record Dates: First submitted 2022-03-07; First posted 2022-03-31 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign Prostatic Hyperplasia; High freqnence Irreversible electroporation; Trans Urethral Resection Prostate
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High Freqnence Irreversible Electroporation (Experimental): Using high freqnence irreversible electroporation to treat patients with benign prostatic hyperplasia
  Interventions: Procedure: High freqnence Irreversible electroporation
- Trans Urethral Resection Prostate (Active Comparator): Using trans urethral resection prostate to treat patients with benign prostatic hyperplasia
  Interventions: Procedure: Trans Urethral Resection Prostate

INTERVENTIONS:
Procedure: High freqnence Irreversible electroporation — High freqnence Irreversible electroporation will be performed via the perineum with the guidance of ultrasound under general anaesthesia to the patient with benign prostatic hyperplasia
  Arms: High Freqnence Irreversible Electroporation
Procedure: Trans Urethral Resection Prostate — Trans urethral resection prostate will be performed under general anaesthesia to the patient with benign prostatic
  Arms: Trans Urethral Resection Prostate

SUMMARY:
This trial is comparing the effects and safety in treating men with benign prostatic hyperplasia between high freqnence irreversible electroporation and trans urethral resection prostate.

DETAILED DESCRIPTION:
A Prospective, Single-center, Randomized Controlled Trial Comparing the Efficacy and Safety of High-Frequency Irreversible Electroporation and Trans Urethral Resection Prostate for Benign Prostatic Hyperplasia

One hundred and seventy-six patients with benign prostatic hyperplasia will include in this study. The clinical trial validation process will be as follows: (1) all patients are randomly divided into two arms: arm 1, high-freqnence irreversible electroporation; arm 2, transurethral resection prostate. The primary outcome is the change in maximum urinary flow rate and urinary symptoms by questionnaire of International Prostate Symptom Score at 3 months after surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 40 years old
2. IPSS>8
3. Qmax <15ml/s
4. Prostatic volume range of 30 to 100ml, measured by MRI
5. Fully understand the clinical trial protocol and sign the informed consent

Exclusion Criteria:

Have a history of prostate cancer or patients suspicious of prostate cancer Neurogenic bladder Metal implants in their body Previous history of prostatic or urethral surgery With Catheterisation more than 2 weeks Any other conditions that investigator judges that participations who are not suitable for this trial

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 118 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
maximum urinary flow rate(Qmax) | 1 and 3 months after surgical treatment
  the change from baseline in maximum urinary flow rate(Qmax)
urination function(evaluated by International prostate symptom score, IPSS) | 1 and 3 months after surgical treatment
  the change from baseline in IPSS (International prostate symptom score)

SECONDARY OUTCOMES:
sexual function evaluated by International Index of Erectile Function Questionnaire-5 (IIEF-5) | 1 and 3 months after surgical treatment
  the change from baseline in International Index of Erectile Function Questionnaire-5 (IIEF-5)
sexual function evaluated by the International Consultation on Incontinence Questionnaire Male Sexual Matters Associated with Lower Urinary Tract Symptoms Module (ICIQ--MLUTSsex) | 1 and 3 months after surgical treatment
  the change from baseline in International Consultation on Incontinence Questionnaire Male Sexual Matters Associated with Lower Urinary Tract Symptoms Module (ICIQ--MLUTSsex)
post-void residual urine volume (PVRU) | 1 and 3 months after surgical treatment
  the change from the baseline in the post-void residual urine volume (PVRU)
urinary incontinence evaluated by ICIQ (International Consultation on Incontinence Questionnaire) | 1 and 3 months after surgical treatment
  the change from baseline in by ICIQ (International Consultation on Incontinence Questionnaire)
urinary incontinence evaluated by separate EPIC (Expanded Prostate Cancer Index Composite) pad-use item | 1 and 3 months after surgical treatment
  the change from the baseline in urinary incontinence, evaluated by separate EPIC (Expanded Prostate Cancer Index Composite) pad-use item
quality of life (QOL) evaluated by IPSS QoL subscore | 1 and 3 months after surgical treatment
  the change from the baseline in QOL, evaluated by IPSS QoL subscore
quality of life (QOL) evaluated by Hospital Anxiety and Depression Scale (HADS)) | 1 and 3 months after surgical treatment
  the change from the baseline in QOL, evaluated by Hospital Anxiety and Depression Scale (HADS)
perioperative parameters(operative time) | 1 month
  operative time
perioperative parameters(the postoperative hospital stay) | 1 month
  the postoperative hospital stay
perioperative parameters(haemoglobin declination) | 6 hours, 24 hours after surgical treatment
  haemoglobin declination
perioperative parameters(serum sodium declination) | 6 hours, 24 hours after surgical treatment
  serum sodium declination
perioperative parameters(catheterisation duration) | 1 month
  catheterisation duration
early postoperative urinary symptoms | 1 and 3 months after surgical treatment
  include dysuria, urgency, or post micturition pain
pain measured by a surgical pain scale | 24 hours, 1 week, 1 month and 3 months
  pain measured by a surgical pain scale range from 0 to 10
adverse event | 1 and 3 months after surgical treatment
  including TUR syndrome, blood transfusion, clot retention, uti, transient incontience, retrograde ejaculation.
voided volume | 1 and 3 months after surgical treatment
  the change from the baseline in voided volume

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Wang, Principal Investigator — Shanghai East Hospital,Tongji University School of Medicine
Locations (1):
- Haifeng Wang, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication will be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and supporting information will be available after the first relevant article is published and last for 10 years after the latest relevant article is published.
Access Criteria: Approvals need to be sort from the data custodians at the health services involved in line with China regulations

REFERENCES:
- [Derived] He BM, Shi ZK, Chen R, Wang HF. Study protocol for a single-centre non-inferior double-blinded randomised controlled trial in China comparing the efficacy and safety of high-frequency irreversible electroporation with transurethral resection of the prostate in treating lower urinary tract symptoms and benign prostatic obstruction (the GIANT trial). BMJ Open. 2025 Jan 9;15(1):e092489. doi: 10.1136/bmjopen-2024-092489. PMID 39788775